CLINICAL TRIAL: NCT05695209
Title: Equity Using Interventions for Pain and Depression (EQUIPD) - Phase 1
Brief Title: Equity Using Interventions for Pain and Depression - Pilot Study
Acronym: EQUIPD-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Marianne S. Matthias, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16571; R61NR020845 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Depression; Health Equity
Keywords: chronic pain; depression; health equity; shared decision making; decision aid
MeSH Terms: conditions — Chronic Pain; Depression | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching and Decision Aid (Experimental): Individual coaching sessions and Decision Aid
  Interventions: Behavioral: Coaching and Decision Aid
- Control (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: Coaching and Decision Aid — Four (4) coaching sessions over approximately 12 weeks with integration of Decision Aid contents
  Arms: Coaching and Decision Aid

SUMMARY:
This project is part of the NIH Helping to End Addiction Long-term (HEAL) initiative (https://heal.nih.gov/). This pilot randomized controlled trial (RCT) is part of phase 1 of a two-phase, 5-year project with the overarching goal of testing a decision aid (DA)/coaching intervention, tailored to Black patients with comorbid chronic pain and depression, to encourage use of and adherence to nonpharmacological pain treatments (NPTs).

This 2-arm pilot trial randomized 30 Black patients with comorbid chronic musculoskeletal pain and depression in primary care from an urban safety-net health system. After the baseline assessment, patients randomized to the intervention were asked to participate in 4 coaching sessions over approximately 12 weeks. Sessions used Motivational Interviewing principles to foster openness to NPTs and self-efficacy by helping patients identify their goals and priorities, understand their NPT options, prepare them to discuss and choose options with their primary care providers (PCPs), and reinforce these choices to foster maintenance of these changes. DA contents were integrated into these sessions, which facilitated discussion of these options with their PCP. The first 3 sessions ideally took place prior to the patient's next scheduled PCP visit; the final session occurred after this visit. Assessments were conducted at baseline, 3 months (i.e., after completing the final coaching session), and 6 months.

Patients randomized to the wait-list control group received usual care (in addition to study assessments at baseline, 3 months, and 6 months). After completing the final assessment, they were given the DA and offered a 20-minute coaching session to walk them through it (patients could decline the coaching session).

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must:

* have musculoskeletal pain in the low back, cervical spine, or extremities (hip, knee, shoulder) for ≥3 months,
* have at least moderate pain intensity and interference with function, defined by a score ≥4 (possible range: 0-10) on the Pain, Enjoyment of Life and General Activity scale (PEG), a 3-item measure of pain intensity, interference with enjoyment of life, and interference with general activity,
* have at least mild depression, defined as PHQ-8 score ≥5,
* identify as Black or African American,
* have consistent access to a telephone,
* indicate openness to new pain treatments, and
* have a scheduled appointment with their PCP in the next approximate 2-4 months

Exclusion Criteria:

Patients are excluded:

* if previously participated in the PI's past pilot study (IRB #12885) or participation as a Patient Engagement Panel member for this project,
* if medical records indicate severe medical conditions likely precluding participation (e.g., NY Heart Association Class III or IV heart failure), or
* if the eligibility screener reveals (1) active suicidal ideation, or (2) severe hearing/speech or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Matthias, PhD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health Primary Care, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH intends to maximize the impact of HEAL Initiative-supported projects through broad and rapid data sharing. All HEAL Initiative award recipients, regardless of the amount of direct costs requested for any one year, are required to comply with the HEAL Public Access and Data Sharing Policy, which also aligns with the NIH Policy for Data Management and Sharing (https://grants.nih.gov/grants/guide/notice-files/NOT-OD-21-013.html). HEAL award recipients must following all requirements and timelines developed through the HEAL Initiative Data Ecosystem, as described in HEAL's compliance guidance (https://heal.nih.gov/data/complying-heal-data-sharing-policy).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication of the primary manuscript
Access Criteria: Implementation of the plan will follow the HEAL Public Access and Data Sharing Policy.
URL: https://heal.nih.gov/data/public-access-data

REFERENCES:
- Available data/document: Individual Participant Data Set: VIV00009027 — https://vivli.org — https://doi.org/10.25934/PR00009027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible participants (primary care patients within an academic, safety-net healthcare system) were identified through electronic medical records and sent a letter and brochure describing the study. A study team member followed up with a phone call to assess interest and, if interested, screen for eligibility.
Period: 3-months
Arm/Group | Coaching and Decision Aid | Control
Started | 16 | 14
Completed | 14 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Unable to contact for 3-month data collection | 0 | 1
Period: 6-months
Arm/Group | Coaching and Decision Aid | Control
Started | 14 | 14 (We attempted to collect data from all non-withdrawn participants. We were unable to contact 1 participant for 3-month data collection; however, we were able to collect 6-month data from that participant. A different participant was lost to follow-up at 6 months.)
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coaching and Decision Aid | Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (14.3) | 61.3 (13.4) | 60.6 (13.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 5 | 9
  Female | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 14 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 0 | 0 | 0
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Highest level of education completed [Count of Participants; unit: Participants]
  Some Secondary School or High School Education | 5 | 1 | 6
  High School (or Secondary School) Degree Complete | 7 | 5 | 12
  Associate's or Technical Degree Complete | 4 | 5 | 9
  College/Baccalaureate/Doctoral or Postgraduate Education | 0 | 3 | 3
Current relationship status [Count of Participants; unit: Participants]
  Divorced/Separated | 3 | 7 | 10
  Married/Domestic Partner | 2 | 1 | 3
  Never Married | 8 | 2 | 10
  Widowed | 2 | 4 | 6
  Other | 1 | 0 | 1
Employment status [Count of Participants; unit: Participants]
  Full-time employment | 2 | 4 | 6
  Not employed | 13 | 7 | 20
  Part-time employment | 1 | 3 | 4
Household income [Count of Participants; unit: Participants] — When you consider your household income from all sources (today), would you say that you are comfortable, have just enough to makes ends meet, or do not have enough to make ends meet?
  Participants
    Comfortable | 2 | 2 | 4
    Just enough to make ends meet | 10 | 8 | 18
    Not enough to make ends meet | 4 | 4 | 8
Pain duration [Mean (Standard Deviation); unit: months] — How long (months) have you had the type of pain for which you are enrolled in this study?
  months | 140.6 (117.2) | 146.2 (165.9) | 143.2 (139.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Brief Pain Inventory (BPI) Interference Scale at 3 Months
Description: The pain interference score averages seven ratings, 0 (does not interfere) to 10 (interferes completely), of interference with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 14 | 13
units on a scale | -1.02 (1.87) | -0.30 (2.24)

2. Primary Outcome: Change From Baseline Brief Pain Inventory (BPI) Interference Scale at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 12
units on a scale | -1.75 (2.28) | -1.14 (1.51)

3. Secondary Outcome: Change From Baseline Patient Health Questionnaire (PHQ)-8 at 3 Months
Description: The PHQ-8 is a widely-used, validated 8-item measure of depression severity. The PHQ-8 is scored by assigning a value of 0 (not at all) to 3 (nearly every day) to each of the 8 items, with a total score ranging from 0 to 24. Higher scores indicate worse depression severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 14 | 13
units on a scale | -2.36 (5.57) | -0.77 (4.44)

4. Secondary Outcome: Change From Baseline Patient Health Questionnaire (PHQ)-8 at 6 Months
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | -2.15 (4.18) | -0.46 (4.75)

5. Secondary Outcome: Change From Baseline Generalized Anxiety Disorder Scale (GAD-7) at 3 Months
Description: Anxiety will be measured with the 7 item Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 is scored by assigning a value of 0 to 3 to each of the seven items, with a total score ranging from 0 to 21. The total score indicates the severity of anxiety symptoms (higher scores indicating a worse outcome).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 14 | 13
units on a scale | -3.29 (5.01) | -0.08 (6.30)

6. Secondary Outcome: Change From Baseline Generalized Anxiety Disorder Scale (GAD-7) at 6 Months
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | -3.23 (3.75) | -0.23 (4.40)

7. Secondary Outcome: Change From Baseline Pain Catastrophizing Scale at 3 Months
Description: The Pain Catastrophizing Scale is a 13-item scale that assesses catastrophizing-a cognitive-emotional factor that predicts poor treatment response. The scale uses a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time) for each item with a total score ranging from 0 to 52. Higher scores indicate a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | -4.31 (11.26) | 3.54 (8.78)

8. Secondary Outcome: Change From Baseline Pain Catastrophizing Scale at 6 Months
Description: as for outcome 7
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | -5.00 (13.39) | -2.12 (12.01)

9. Secondary Outcome: Change From Baseline Altarum Consumer Engagement (ACE) Measure at 3 Months
Description: Patient engagement will be measured with the 12-item Altarum Consumer Engagement (ACE) Measure, which has 3 subscales: 1) commitment to manage one's health, 2) informed choice, and 3) confidence to participate in treatment decisions. Each item is assessed on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree) with a total score ranging from 0 to 48. Higher scores indicate greater engagement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 2.64 (8.96) | -2.04 (9.16)

10. Secondary Outcome: Change From Baseline Altarum Consumer Engagement (ACE) Measure at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 4.29 (7.16) | -0.24 (10.93)

11. Secondary Outcome: Change From Baseline Use of Nonpharmacological and Self-Care Approaches (NSCAP) at 3 Months
Description: The NSCAP asks about 9 nonpharmacological treatment (NPT) modalities and assesses details of use such as frequency, location/source of service, and patients' judgments of effectiveness. Space is also provided for other NPTs that are used but not listed. The number of modalities for which patients answer "yes" will be summed for analyses.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: counts of NPTs
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
counts of NPTs | 0.23 (1.96) | -0.46 (1.61)

12. Secondary Outcome: Change From Baseline Use of Nonpharmacological and Self-Care Approaches (NSCAP) at 6 Months
Description: as for outcome 11
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: counts of NPTs
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
counts of NPTs | 0.38 (1.50) | 0.54 (1.94)

13. Secondary Outcome: Change From Baseline Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) at 3 Months
Description: Communication self-efficacy will be measured with this 5-item scale that measures patients' self-efficacy in obtaining medical information and getting their most important health concern discussed in a clinic visit. Higher scores indicate greater communication self-efficacy. The scale uses ratings from 0 (not at all confident) to 10 (extremely confident) for each item with a total score ranging from 0 to 50.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
score on a scale | 0.08 (5.45) | 2.08 (10.90)

14. Secondary Outcome: Change From Baseline Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) at 6 Months
Description: as for outcome 13
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 1.46 (4.41) | 0.15 (8.71)

15. Secondary Outcome: Change From Baseline CollaboRATE at 3 Months
Description: Shared decision making will be measured with CollaboRATE, a 3-item measure assessing provider effort from the patient's perspective to engage in shared-decision making during a recent appointment. The CollaboRATE scale uses a 5-point Likert scale, ranging from "No effort was made (0)" to "Every effort was made (4)" for each item with a total score ranging from 0 to 12. Higher scores indicate higher provider effort from the patient's perspective to engage in shared-decision making.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 0.26 (0.47) | -0.13 (0.91)

16. Secondary Outcome: Change From Baseline CollaboRATE at 6 Months
Description: Shared decision making will be measured with CollaboRATE, a 3-item measure assessing provider effort from the patient's perspective to engage in shared-decision making during a recent appointment. The CollaboRATE scale uses a 5-point Likert scale, ranging from "No effort was made (0)" to "Every effort was made (4)" or each item with a total score ranging from 0 to 12. Higher scores indicate higher provider effort from the patient's perspective to engage in shared-decision making.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 0.26 (0.71) | -0.05 (0.49)

17. Secondary Outcome: Change From Baseline Working Alliance Inventory (WAI) Client Short Form at 3 Months
Description: The Working Alliance Inventory (WAI) Client Short Form assesses patient-provider agreement on treatment goals, collaboration to achieve these goals, and degree of emotional bond (liking and trust) between patients and providers. The scale uses ratings from 1 (Never) to 7 (Always) for each item with a total score ranging from 12 to 84. Higher scores indicate greater alliance between patient and provider.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 3.67 (13.34) | -5.54 (13.08)

18. Secondary Outcome: Change From Baseline Working Alliance Inventory (WAI) Client Short Form at 6 Months
Description: The Working Alliance Inventory (WAI) Client Short Form assesses patient-provider agreement on treatment goals, collaboration to achieve these goals, and degree of emotional bond (liking and trust) between patients and providers. The scale uses ratings from 1 (Never) to 7 (Always) or each item with a total score ranging from 12 to 84. Higher scores indicate greater alliance between patient and provider.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Decision Aid | Control
Number analyzed (Participants) | 13 | 13
units on a scale | 5.69 (9.78) | -2.38 (8.05)

ADVERSE EVENTS:
Time Frame: approximately 6 months
Description: Adverse events were not systematically collected for this study that was determined to be minimal risk by the Institutional Review Board.
Groups:
- Control: Received Decision Aid: Wait-list control group
- Control: Usual Care Without Decision Aid: Control, did not receive Decision Aid
Arm/Group | Coaching and Decision Aid | Control: Received Decision Aid | Control: Usual Care Without Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05695209/Prot_001.pdf
  • Statistical Analysis Plan (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT05695209/SAP_002.pdf
  • Informed Consent Form (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT05695209/ICF_003.pdf